CLINICAL TRIAL: NCT04881240
Title: A Phase I Study Evaluating Allogeneic Memory T Cells Engineered to Express Chimeric Antigen Receptors Specific for CD19 for the Treatment of Pediatric and Young Adult Patients ≤ 21 Years of Age With Relapsed or Refractory CD19-Positive Leukemia
Brief Title: Study of CD19-directed Allogeneic Memory T-cell Therapy for Relapsed/Refractory CD19+ Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEMCAR19
Record Dates: First submitted 2021-04-27; First posted 2021-05-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia, Refractory; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Mesna; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Participants in group A have received a prior stem cell transplant from their CAR T-cell donor.
  Interventions: Biological: CD19-CAR(Mem) T-cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Device: CliniMACS; Procedure: Leukapheresis
- Group B (Experimental): Participants in group B have not received a prior stem cell transplant from their CAR T-cell donor.
  Interventions: Biological: CD19-CAR(Mem) T-cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Device: CliniMACS; Procedure: Leukapheresis

INTERVENTIONS:
Biological: CD19-CAR(Mem) T-cells — Allogeneic CD19-CAR.CD45RA-negative T-cells Intravenous infusion
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard derivative. It acts as an alkylating agent that causes cross-linking of DNA strands by binding with nucleic acids and other intracellular structures, thus interfering with the normal function of DNA.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine phosphate is a synthetic purine nucleoside analog. It acts by inhibiting DNA polymerase, ribonucleotide reductase and DNA primase by competing with the physiologic substrate, deoxyadenosine triphosphate, resulting in inhibition of DNA synthesis.
  Other Names: Fludara
Drug: Mesna — Mesna is a synthetic sulfhydryl (thiol) compound. Mesna contains free sulfhydryl groups that interact chemically with urotoxic metabolites of oxaza-phosphorine derivatives such as cyclophosphamide and ifosfamide.
  Other Names: Mesnex
Device: CliniMACS — A CliniMACS device is used to select donor T-cells for manufacturing of the memory CAR T-cell product.
Procedure: Leukapheresis — Leukapheresis is performed to collect the T cells that are needed to generate the CD19-CAR.CD45RA-negative T-cells product for the clinic study.

SUMMARY:
This is a Phase I clinical study evaluating the safety and maximum tolerated dose of a novel CAR T-cell product: allogeneic memory (CD45RA- negative) T-cells expressing a CD19-specific CAR 41BBz (CD19-CAR.CD45RA- negative T-cells) for the treatment of patients ≤ 21 years old with relapsed and/ or refractory CD19-positive leukemia.

Primary Objective

To determine the maximum tolerated dose (MTD) and characterize the safety profile and dose-limiting toxicities (DLTs) of treatment with allogeneic CD19-CAR.CD45RA-negative T-cells in pediatric, adolescent and young adult patients ≤ 21 years of age, with relapsed and/or refractory CD19-positive leukemia.

Secondary Objectives

* To evaluate the anti-leukemic activity of allogeneic CD19-CAR.CD45RA-negative T-cells.
* To determine rates and severity of graft-versus-host-disease (GVHD) after treatment with allogeneic CD19-CAR.CD45RA-negative T-cells.

Exploratory Objectives

* To study the expansion, persistence and phenotype of allogeneic CD19-CAR.CD45RA-negative T-cells.
* To characterize the cytokine profile in the peripheral blood and CSF after treatment with allogeneic CD19-CAR.CD45RA-negative T-cells.
* To assess whether allogeneic CD19-CAR.CD45RA-negative T-cells acquire functional versus exhaustion-associated epigenetic programs.
* To determine immune reconstitution post treatment, and the clonal structure and endogenous repertoire of allogeneic CD19-CAR.CD45RA-negative T-cells and relate inferred specificity to CAR response profiles.
* To characterize incidence and mechanisms of relapse post-therapy with allogeneic CD19-CAR.CD45RA-negative T-cells.

DETAILED DESCRIPTION:
This is a Phase I dose escalation study using a 3+3 study design. Two groups of patients will be evaluated in this study: group A - patients have received a prior stem cell transplant from their CAR T-cell donor; group B - patients have not received a prior stem cell transplant from their CAR T-cell donor. There will be up to 30 participants per group and a donor/ family member for each patient.

.

ELIGIBILITY:
Inclusion Criteria Eligibility Criteria for Donors: Apheresis and Manufacturing

* Age ≥ 18 years old
* At least single haplotype matched (≥ 3/6) family member
* HIV negative
* For females of child bearing age: Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment AND Not lactating with intent to breastfeed
* Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance

For Cohort A only, identified recipient with relapsed and/or refractory CD19-positive leukemia

For Cohort B only, iIdentified recipient with relapsed and/or refractory CD19-positive leukemia who is not suitable to receive autologous CD19-CAR T-cell therapy as defined by the following:

* Relapsed and/or refractory disease despite prior treatment with autologous CD19- CAR T-cell therapy
* History of prior autologous leukapheresis failure
* History of prior autologous CAR T-cell manufacturing failure
* Unable to undergo autologous leukapheresis in the opinion of the study PI(s): examples may include - patient small size/low weight, inadequate T-cell counts, rapidly progressive leukemia, clinical status not amenable to apheresis

Eligibility Criteria for Patients: Treatment

* Age ≤ 21 years old
* Relapsed and/or refractory CD19-positive leukemia*:

  * Refractory disease (defined as any of the following):

    * Primary refractory disease despite at least 2 cycles of an intensive chemotherapy regimen designed to induce remission
    * Refractory disease despite salvage therapy
  * Relapsed disease (defined as any of the following):

    * 2nd or greater relapse
    * Any relapse after allogeneic hematopoietic cell transplantation (HCT)
    * 1st relapse if patient requires an allogeneic HCT as part of standard of care relapse therapy, but is found to be ineligible and/or unsuitable for HCT

CD19-positivity confirmed within 2 months and after receipt of any CD19-directed therapy

* Patient cohorts:

  * Cohort A: patient has previously received a HCT from the selected CAR T-cell donor
  * Cohort B - patient has NOT previously received a HCT from the selected CAR T-cell donor.
* For Cohort B only, not suitable to receive autologous CD19-CAR T-cell therapy as defined above in Criteria: Eligibility Criteria for Donors: Apheresis and Manufacturing
* Detectable medullary CD19-positive leukemia
* Estimated life expectancy of ≥ 8 weeks
* Karnofsky or Lansky performance score ≥ 50
* No CNS-3 disease or any level of detectable leukemia in CNS with associated neurologic symptoms
* If history of allogeneic HCT (regardless of donor type), prior to planned CAR T-cell infusion, must meet the following criteria:

  * ≥ 3 months from HCT
  * have recovered from prior HCT therapy
  * have no evidence of active GVHD within prior 2 months
  * have not received a donor lymphocyte infusion (DLI) within the 28 days prior to planned CAR T-cell infusion
* Adequate cardiac function: left ventricular ejection fraction ≥ 40% or shortening fraction ≥ 25% (function may be supported by pharmacologic therapy)
* EKG without evidence of clinically significant arrhythmia
* Adequate renal function: creatinine clearance or radioisotope GFR 50 ml/min/1.73m2 (GFR 40 ml/min/1.73m2 if < 2 years of age)
* Adequate pulmonary function: forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing
* Total bilirubin ≤ 3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age
* No history of HIV infection
* No evidence of severe, uncontrolled bacterial, viral or fungal infection
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For females of child bearing age:

  * Not pregnant with negative serum or urine pregnancy test ≤ 7 days prior to enrollment AND Not lactating with intent to breastfeed
* If sexually active, agreement to use birth control until 6 months after CAR T-cell infusion
* No history of hypersensitivity reactions to murine protein-containing products
* Not receiving systemic steroids therapy exceeding the equivalent of 0.5 mg/kg/day of methylprednisolone ≤ 7 days prior to CAR T-cell infusion
* Not receiving systemic therapy ≤ 14 days prior to CAR T-cell infusion, which will interfere with the activity of the CAR T-cell product in vivo (in the opinion of the study PI(s))
* Not receiving intrathecal chemotherapy ≤ 7 days prior to CAR T-cell infusion

Exclusion Criteria:

NA

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of allogeneic, CD19-CAR.CD45RA-negative cells | 4 weeks after CAR T-cell infusion
  This phase I study includes dose escalation/de-escalation based on dose limiting toxicity (DLT) assessment to determine the maximum tolerated dose (MTD) of allogeneic, CD19-CAR.CD45RA-negative cells.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee C. Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital; Stephen Gottschalk, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols